CLINICAL TRIAL: NCT05691010
Title: A Feasibility Study of Integrated Delivery of Hypofractionated Pelvic IMRT With Carboplatin and Paclitaxel in Stage III Copy-Number Low and Copy-Number High Subtypes of Endometrial Cancer
Brief Title: A Study of Short-Course Radiation Therapy With Chemotherapy in People With Endometrial Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-405
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer; Stage III Endometrial Cancer; Stage III Endometrial Carcinoma; Endometrial Carcinoma; Endometrial Carcinoma Stage III
Keywords: endometrial cancer; endometrial cancer stage III; endometrial carcinoma stage III; stage III endometrial cancer; stage III endometrial carcinoma; Memorial Sloan Kettering Cancer Center; 22-405
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Endometrial Cancer (Experimental): Participants have stage III endometrial cancer
  Interventions: Radiation: Intensity-modulated radiation therapy; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy — After cycles 1, 2, 3 or 4 of chemotherapy, patients will receive IMRT to the vaginal cuff and pelvic lymph nodes with a total dose of 25 Gy delivered in 5 daily fractions of 5 Gy
  Other Names: IMRT
Drug: Carboplatin — Patients enrolled in this trial will receive chemotherapy with carboplatin IV AUC 5 at the discretion of the treating investigator plus paclitaxel 175 mg/m2 every 21 days for 6 cycles
Drug: Paclitaxel — Patients enrolled in this trial will receive chemotherapy with carboplatin IV AUC 5 at the discretion of the treating investigator plus paclitaxel 175 mg/m2 every 21 days for 6 cycles

SUMMARY:
The purpose of this study is to find out whether short-course radiation therapy (1 week instead of the usual 5 weeks) with chemotherapy (carboplatin and paclitaxel) is practical (feasible), meaning that most participants are able to complete the treatment schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed endometrial carcinoma. The following histologic subtypes are eligible for inclusion: endometrioid, serous, clear cell, dedifferentiated/undifferentiated, mixed epithelial, adenocarcinoma not otherwise specified, and carcinosarcoma.
* Surgery must have included a hysterectomy, bilateral salpingo-oophorectomy, and pelvic lymph node surgical assessment (sentinel lymph node mapping and/or sampling). Para-aortic lymph node surgical assessment is optional.
* Patients must have FIGO (2009) stage IIIA or IIIC1 disease (as determined by surgical staging).
* Patients must consent to testing with MSK-IMPACT part A and are encouraged to consent to both parts A and C.
* Age ≥ 18 years.
* Patients must have an Karnofsky Performance Status (KPS) ≥ 70 (or ECOG 0 or 1).
* Neurologic function: Neuropathy (sensory and motor) grade ≤ 1.
* No residual gross disease after surgery.
* No prior radiation therapy or chemotherapy for treatment of endometrial cancer.
* No active infection requiring antibiotics, except for uncomplicated urinary tract infection.
* Patients must have adequate organ function, defined by the following laboratory results no more than 14 days prior to first study treatment:

  * Absolute neutrophil count (ANC) ≥ 1500/mcL
  * Platelet count ≥ 100,000/mcL
  * AST/ALT ≤ 3X upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5X ULN. Patients with known Gilbert's disease and a total bilirubin ≤ 3X ULN may be enrolled.
  * Creatinine ≤ 1.5X ULN
* Entry into study is limited to no more than 12 weeks from the date of surgery.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients of childbearing age will by definition have undergone hysterectomy and bilateral oophorectomy prior to study enrollment.
* Participants must agree not to breastfeed during the study or for 150 days after the last dose of study treatment.

Exclusion Criteria:

* Patients whose endometrial cancers harbor known pathogenic POLE mutations
* Patients whose endometrial cancers are mismatch repair deficient, as determined by immunohistochemical staining for MLH1, PMS2, MSH2, and MSH6 and/or MSI-H
* Active inflammatory bowel disease, such as Crohn's disease or ulcerative colitis.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. This includes but is not limited to: uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, and superior vena cava syndrome.
* Patients unfit for pelvic radiation therapy due to the following:

  * Has had radiation therapy encompassing >20% of the bone marrow within 2 weeks, or any radiation therapy within 1 week prior to day 1 of protocol therapy
  * Patients with a history of pelvic radiation.
  * Patients with a history or current diagnosis of a vesicovaginal, enterovaginal, or colovaginal fistula.
  * Any hematological abnormality or disorder that would be a contraindication to radiation per the treating physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of integrated delivery of short-course IMRT with carboplatin/paclitaxel in patients with stage III endometrial cancer | up to 3 years
  Feasibility of study treatment is defined as defined as the number of participants who complete all 6 planned cycles of carboplatin and paclitaxel with no delays in chemotherapy cycles greater than 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Kaled Alektair, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org